CLINICAL TRIAL: NCT06469398
Title: A Post Market Study of a Laser System for the Treatment of Acne Vulgaris
Brief Title: A Post Market Device Study for the Treatment of Acne
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-22-AC05
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Laser Treatment (Experimental)
  Interventions: Device: Cutera Laser System

INTERVENTIONS:
Device: Cutera Laser System — Subjects will receive up to 6 laser treatments

SUMMARY:
To evaluate the safety and efficacy of the Cutera laser system for the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male, Fitzpatrick Skin Types I-VI, 16 to 60 years of age (inclusive).
2. Has clinically diagnosed acne vulgaris of severity grade 3 - 4 (moderate to severe) on the face based on photographic review by expert dermatologist grader(s) using the Investigator's Global Assessment Scale.
3. Has ≥ 10 inflammatory acne lesions on the face as determined by the Investigator (or qualified designee).
4. Subject (and parent or legal guardian if subject is a minor under age 18) must be able to read, speak, and understand English and sign the Informed Consent Form.
5. Willing and able to adhere to the treatment and follow-up schedule and pre/post-treatment care instructions.
6. Willing to have very limited sun exposure (including avoiding tanning booths, sun lamps, sunbathing) and use an investigator approved sunblock or sunscreen of SPF 30 or higher on the face every day for the duration of the study, including the follow-up period.
7. Must maintain the same acne treatment regimen, including topical and systemic medications for at least 2 weeks prior to enrollment, and for the duration of the study, including the follow-up period unless approved by the Investigator.
8. Willing to have photographs taken of the face and agree to the use of photographs for presentation, educational or marketing purposes.
9. Agree to not undergo any other procedure(s) or add any new treatment modalities in the target area during the study unless approved by Investigator.
10. Willing to use investigator approved skincare topicals and follow investigator approved skincare regimen for the duration of the study.

Exclusion Criteria:

1. Has clinically diagnosed acne vulgaris of severity grade 0, 1, 2 (clear, almost clear, mild) on the face based on photographic review by expert dermatologist grader(s) using the Investigator's Global Assessment Scale.
2. Prior treatment to the target area during participation in a clinical trial of another device or drug within 1 month (30 days) prior to study participation.
3. Still healing from another treatment in the target area according to investigator's discretion.
4. Currently pregnant or planning on becoming pregnant anytime during the duration of the study.
5. Excessive facial hair (e.g., beards, sideburns, moustaches, etc.) that may preclude treatments, photos, or accurate acne lesion assessments in the target area.
6. Currently undergoing treatment for skin cancer in the target area or undergoing systemic chemotherapy for the treatment of cancer.
7. As per the Investigator's discretion, any physical, mental or medical condition which might make it unsafe for the subject to participate in this study or might interfere with patient's participation in the full study protocol.
8. Known hypersensitivity to, history of allergic reaction to, or contraindication to Pro-Nox or mild oral anti-anxiety or pain medication, if administered.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-18 (Estimated)

PRIMARY OUTCOMES:
Percent of Subjects Who are Responders | 12 weeks post final treatment
  The primary outcome measure to evaluate the efficacy of the Cutera device is the percent of subjects who are responders at 12 weeks post final treatment, where a responder is defined as ≥ 1-point reduction on the Investigator's Global Assessment scale at follow up compared to baseline.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dermatology of Boca, Boca Raton, Florida
  - Schweiger Dermatology PC, Reseach Division, Hackensack, New Jersey
  - Bellaire Dermatology Associates, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No